CLINICAL TRIAL: NCT06737250
Title: Open, Single Arm, Multicenter, Phase 2 Trial to Evaluate Efficacy and Safety of NB02 (Poseltinib) Combined with Rituximab and Lenalidomide As a Salvage Therapy for Patients with Relapsed or Refractory Primary Central Nervous System Lymphoma
Brief Title: NB02 (Poseltinib) Combined Rituximab and Lenalidomide in R/R PCNSL
Acronym: POTENTIAL-P
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NOBO Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240084640
Record Dates: First submitted 2024-12-06; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Primary CNS Lymphoma (PCNSL)
Keywords: Refractory; Relapsed
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: This clinical study is conducted as an open, single-arm study targeting a patient population with rare diseases for which there is no distinct standard of care treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NB02 (Poseltinib) combined Rituximab and Lenalidomide (Experimental)
  Interventions: Drug: R2P -> RP

INTERVENTIONS:
Drug: R2P -> RP — Induction(R2P) 21 days per cycles, 6 cycles
  * NB02 : 60mg BID PO, Day 1-21
  * Rituximab 375mg/m2 DAY IV Day 1, 8, 15 at 1st cycle; D1 at 2nd to 6th cycles
  * Lenalidomide : 20mg QD PO, Day 1-14
  Maintenance(RP) 21 days per cycles, until Progression
  * NB02 : 60mg BID PO, Day 1-21
  * Lenalidomide : 20mg QD PO, Day 1-14

SUMMARY:
An Open, Single treatment arm, Multi-center, Prospective, Phase 2 Trial to Evaluate Efficacy and Safety of NB02 (Poseltinib) combined with Rituximab and Lenalidomide as a Salvage Therapy for Patients with Relapsed or Refractory Primary Central Nervous System Lymphoma

DETAILED DESCRIPTION:
For outpatients or inpatients who meet the criteria for subject selection, the study is conducted with patients who have given a sufficient explanation of the study and who voluntarily consented to participate in the study.

Patients enrolled in the study receive a combination therapy of NB02, Rituximab and lenalidomide according to the criteria specified in the protocol.

Induction(R2P) 21 days per cycles, 6 cycles

* NB02 : 60mg BID PO, Day 1-21
* Rituximab 375mg/m2 DAY IV Day 1, 8, 15 at 1st cycle; D1 at 2nd to 6th cycles
* Lenalidomide : 20mg QD PO, Day 1-14

Maintenance(RP) 21 days per cycles, until Progression

* NB02 : 60mg BID PO, Day 1-21
* Lenalidomide : 20mg QD PO, Day 1-14

ELIGIBILITY:
Inclusion Criteria:

1. A patient who voluntarily decided to participate and provided written consent after receiving an explanation of this clinical trial and the characteristics of the investigational drug.
2. Adults aged 19 years or older and 80 years or younger.
3. Patients diagnosed histopathologically with CD20-positive primary central nervous system lymphoma (PCNSL).
4. Patients with confirmed disease progression or treatment resistance after remission induction therapy, radiotherapy, or autologous transplantation, with no more than two prior systemic treatments and no more than one prior radiotherapy treatment (preconditioning and transplantation for hematopoietic stem cells are counted as one systemic treatment; radiotherapy, regardless of fractionation or dose, including concurrent chemoradiotherapy, is counted as one treatment).
5. Patients with measurable lesions identified by gadolinium-enhanced brain MRI (CT may be used if MRI is contraindicated).
6. Patients with an ECOG Performance Status (PS) score of 2 or less.
7. Patients who agree to comply with the Pregnancy Prevention Plan (PPP) for lenalidomide.
8. Patients with an expected survival of at least 3 months, as judged by the investigator.

Exclusion Criteria:

1. Patients newly diagnosed with primary central nervous system lymphoma (PCNSL).
2. Patients with ocular lymphoma without brain lesions.
3. Patients with metastatic CNS lymphoma involving organs outside the central nervous system, except th eeyes and cerebrospinal fluid (if systemic disease is present: Secondary CNS lymphoma).
4. Patients whose screening laboratory test results meet the following criteria (⁕ corrected after transfusion or use of hematopoietic growth factors are acceptable):

(1) Absolute neutrophil count <1,000/μL (at least 2 weeks after G-CSF administration).

(2) Platelet count <75,000/μL (at least 1 week after platelet transfusion). (3) Hemoglobin <9.0 g/dL (at least 2 weeks after red blood cell transfusion). (4) Serum calcium >12.0 mg/dL. (5) Serum creatinine >1.5 x the upper normal limit (UNL) or creatinine clearance <60 mL/min (based on the Cockcroft-Gault formula).

(6) Alanine aminotransferase (ALT) >3 × UNL. (7) Aspartate aminotransferase (AST) >3 × UNL. (8) Total bilirubin >1.5 × UNL (Gilbert syndrome: up to 3 × UNL).

* Patients with cardiovascular, hepatic, renal, neurological, immune, infectious, or psychiatric disorders that could affect safety, trial evaluation, or protocol compliance (e.g., regular visits).

  5. The following heart conditions:
  1. Symptomatic or uncontrolled angina and congestive heart failure.
  2. Arrhythmias requiring medication (controlled cases with medication are allowed).
  3. Clinically significant myocardial infarction within 6 months before trial participation.

  6. History of thrombosis or embolism within 6 months before screening.

  7. Gastrointestinal bleeding above Grade 2 according to CTCAE within 6 months before screening.

  8. Ongoing infection above Grade 2 according to CTCAE at the time of screening.

  9. Severe hepatic impairment (e.g., cirrhosis), chronic hepatitis with HBV reactivation.
  * Patients with HBsAg (-) and HBcAb (-), or HBsAg (-) and HBcAb (+) with undetectable HBV DNA, can participate. Prophylactic antiviral therapy and HBV DNA monitoring (every 3-4 weeks) are required for HBcAb (+) cases with undetectable HBV DNA.

    10. Uncontrolled hepatitis C virus (HCV) infection.
  * Patients with negative HCV antibodies or undetectable HCV RNA can participate with HCV RNA monitoring (every 1 cycle).

    11. HIV infection. Patients with negative HIV antibodies or antigen-negative despite HIV antibody positivity can participate.

    12. Severe renal impairment requiring hemodialysis or hemofiltration at screening.

    13. Known immunodeficiency disorders.

    14. Known autoimmune diseases (e.g., multiple sclerosis, acute disseminated encephalomyelitis, rheumatoid arthritis).

    15. History of severe cutaneous adverse reactions (SCARs), including erythema multiforme, Stevens-Johnson syndrome, toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms (DRESS), or acute generalized exanthematous pustulosis (AGEP).

    16. History of malignancies other than the target disease, except:
    1. No treatment for malignancy and disease-free for at least 5 years before screening.
    2. Completely cured with no evidence of recurrence for malignancies within 5 years if surgically treated (e.g., Stage I/II papillary or follicular thyroid cancer, basal cell/squamous cell carcinoma, cervical dysplasia or carcinoma in situ, early-stage stomach or colorectal cancer).

    17. Patients suspected of moderate dementia (K-MMSE-2 score ≤17).

    18. Patients unable to take oral medication.

    19. Hypersensitivity to study drugs (rituximab, lenalidomide, poseltinib) or excipients.

    20. Prior use of lenalidomide, poseltinib, or other BTK inhibitors.

    21. Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

    22. Women who are pregnant or breastfeeding.

    23. Women of childbearing potential⁕ and male participants with female partners of childbearing potential who do not agree to use two reliable contraceptive methods at least 28 days before administration of the investigational drug, during the trial, during temporary discontinuation, and for 12 months after the last administration. (Complete abstinence from heterosexual intercourse is an exception.)
* Women not of childbearing potential include those who have undergone hysterectomy or bilateral oophorectomy, or those in natural menopause for at least 24 consecutive months for non-disease reasons.

  24. Male participants who do not agree to:
  1. Use condoms during the study, even after vasectomy, during temporary discontinuation, and for 12 months after the last administration.
  2. Avoid sperm/semen donation for 12 months after the study.
  3. Immediately inform investigators if their partner becomes pregnant during the study or within 3 months after the study.

  25. Patients with a history of substance abuse, medical, psychiatric, or social conditions that could interfere with trial participation or results.

  26. Patients unable to understand or comply with trial instructions or with a history of poor adherence to medical treatments.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response (ORR) by IRC | 4 cycles (12 weeks)
  End Of Induction

SECONDARY OUTCOMES:
Overall Response by Investigator (ORR) | 4 cycles (12 weeks)
  End Of Induction
Overall Survival (OS) | through study completion, an estimation of 2 years
  End of Study
Progression Free Survival (PFS) | through study completion, an estimation of 2 years
  End Of Treatment
Event Free Survival (EFS) | through study completion, an estimation of 2 years
  End Of Study
Response Duration | through study completion, an estimation of 2 years
  End Of Treatment
Time To Response | through study completion, an estimation of 2 years
  End Of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yul An, Dr, Study Director — NOBO Medicine
Locations (10):
- South Korea (10):
  - Kosin University Gospel Hospital, Busan
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea National Cancer Center, Ilsan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Catholic univ of Yeouido St Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan